CLINICAL TRIAL: NCT02675296
Title: Regional and Long Term Outcomes of Acute Kidney Injury in England From 2000 to 2015 - A National Database Study
Status: Completed | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr. Nitin Kolhe, Consultant Nephrologist, University Hospitals of Derby and Burton NHS Foundation Trust
Other Study IDs: 1.3
Record Dates: First submitted 2016-01-28; First posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Acute Kidney Injury
Keywords: outcome
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute kidney injury requiring dialysis (AKI-D) has increased considerably over last 15 years. The national rise in incidence of acute kidney injury has several ramifications in terms of cost to the health services resulting not only from cost of therapy but also from the later consequences of AKI from development of chronic kidney disease and cardiovascular disease. Mortality in patients with AKI-D is very high and remains unchanged in the last decade in England. In recent years it is becoming clearer that even the national incidence and case-fatality of AKI is influenced by regional variation. In last three decades, many studies have reported unwarranted variation in a wide range of procedures, from the performance of cesarean section and coronary angiography to the treatment of early prostate cancer, stroke, and the ailments of the chronically ill. In surgical care there is evidence that the variation may be driven by forces other than patient illness and medical appropriateness such as access to care and other socioeconomic factors, provider capacity of the local system, medical malpractice pressure, and distinctly different local practices. Despite the public health burden of AKI-D in England, it is unclear if regional variation exists in AKI-D. Variation in incidence of AKI-D in different region of a country may be influenced by patient and physician demographics of the regions, physician preferences or the nature of the hospital serving the population. To reduce the incidence and case fatality of AKI-D, it is imperative to understand if variations in incidence and case-fatality in AKI-D exists in different regions of the country.

To address this gap in knowledge, the investigators combined national database of hospital admissions and discharge with census data from office of national statistic over a period of fifteen years to determine the trend in change in the regional incidence and case fatality of AKI requiring dialysis in England. The investigators also explored various determinants of the regional variation in the dialysis requiring AKI.

Methods Data source The investigators extracted 2000-2015 data from the Hospital Episode Statistics (HES), a data warehouse containing details of all admissions, outpatient appointments, and A&E attendances at National Health Service (NHS) hospitals in England.

Definitions The investigators identified all cases of AKI by using validated International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) codes in any diagnoses codes, in keeping with the objective of the study. Patients with any of the following codes were included: N17.0 for acute renal failure (ARF) with tubular necrosis, N17.1 for ARF with acute cortical necrosis, N17.2 for ARF with medullary necrosis, N17.8 for other ARF and N17.9 for ARF, unspecified. ARF has been replaced by new terminology, AKI, but due to lack of ICD10 codes for AKI, the investigators used the ICD10 codes for ARF and henceforth, will be referred to as AKI in this study. The investigators also extracted all available secondary diagnosis and up to 24 Office of Population Censuses and Surveys Classification of Interventions and Procedures, 4th revision (OPCS-4) codes. To identify patients with AKI-D, the investigators included OPCS code of X40.3 for hemodialysis or X40.4 for hemofiltration in any of the 25 procedures. Patients with chronic kidney disease stage 5 (CKD-5) starting chronic dialysis and end stage renal disease (ESRD) with ICD-10 code of N18.5 and N18.6 respectively were excluded. The investigators also excluded OPCS-4 codes for Arteriovenous fistula (L74.2) or Arteriovenous graft (L74.3) during the inpatient admission. HES data stratifies patient location into 16 different regions. The geographic regions in England were stratified as per the Office of National Statistic (ONS) into nine regions: North East, North West, Yorkshire and Humber, East Midlands, West Midlands, East of England, London, South East and South West. Patients' in geographical locations outside these nine regions were excluded. Patients who were admitted, but were not discharged during the study period will not be included in the study. The investigators also obtained completed hospital discharges from each region to estimate the effect of hospitalization on AKI-D incidence rates, along with number of nephrology consultants in each region from 2000 to 2015 from Health and Social Care Information Centre (HSCIC) in the annual census of medical and dental staff in the NHS. The investigators will also obtain linkage with ONS and UK Renal Registry (UKRR) for long-term patient and renal outcomes. To obtain population incidence of AKI-D for each region, mid-year population of the region in each year from 2000 to 2015 was obtained from the ONS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AKI as identified by International classification of disease, 10th revision (ICD10) of N17 any of the diagnoses codes.
2. AKI patients with procedure code for hemodialysis or for hemofiltration in any of the 25 procedures codes.

Exclusion Criteria:

1. AKI patients who had CKD stage 5 and end stage renal disease
2. AKI patients with procedure codes for arteriovenous fistula or arteriovenous shunt during the inpatient admission.

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The 2000 to 2015 data was extracted from the Hospital Episode Statistics (HES), a data warehouse containing details of all admissions, outpatient appointments and A&E attendances at NHS hospitals in England. HES collects a detailed record for each 'episode' of admitted patient care delivered in England, either by NHS hospitals, primary care trusts, mental health trusts or delivered in the independent sector but commissioned by the NHS. These data are collected during a patient's time in hospital and stored as a large collection of separate records, one for each period of care, in a secure data warehouse.
Sampling Method: Non-Probability Sample
Enrollment: 54680 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incident of AKI-D patients | 15 years
  The study aims to identify regional variation in incidence of AKI-D in each region of England over 15 year period

SECONDARY OUTCOMES:
Number of deaths in each region. | 10 years
  Patient survival over 10 year period
Number of patients developing end stage renal disease | 10 years
  Renal survival over 10 year period
Case-fatality in AKI-D patients | 15 years
  The study aims to identify regional variation in case-fatality of AKI-D in each region of England over 15 year period

CONTACTS AND LOCATIONS:
Overall Officials: Nitin V Kolhe, MD, Principal Investigator — Derby Teaching Hospital NHS Foundation Trust
Locations (1):
- Derby Hospital NHS Foundation Trust, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data is freely available from HSCIC

REFERENCES:
- [Background] Kolhe NV, Muirhead AW, Wilkes SR, Fluck RJ, Taal MW. National trends in acute kidney injury requiring dialysis in England between 1998 and 2013. Kidney Int. 2015 Nov;88(5):1161-9. doi: 10.1038/ki.2015.234. Epub 2015 Jul 29. PMID 26221750
- [Background] Hsu RK, McCulloch CE, Heung M, Saran R, Shahinian VB, Pavkov ME, Burrows NR, Powe NR, Hsu CY; Centers for Disease Control and Prevention Chronic Kidney Disease Surveillance Team. Exploring Potential Reasons for the Temporal Trend in Dialysis-Requiring AKI in the United States. Clin J Am Soc Nephrol. 2016 Jan 7;11(1):14-20. doi: 10.2215/CJN.04520415. Epub 2015 Dec 18. PMID 26683890
- [Background] Hsu RK, McCulloch CE, Ku E, Dudley RA, Hsu CY. Regional variation in the incidence of dialysis-requiring AKI in the United States. Clin J Am Soc Nephrol. 2013 Sep;8(9):1476-81. doi: 10.2215/CJN.12611212. Epub 2013 Aug 8. PMID 23929923
- [Background] Wald R, McArthur E, Adhikari NK, Bagshaw SM, Burns KE, Garg AX, Harel Z, Kitchlu A, Mazer CD, Nash DM, Scales DC, Silver SA, Ray JG, Friedrich JO. Changing incidence and outcomes following dialysis-requiring acute kidney injury among critically ill adults: a population-based cohort study. Am J Kidney Dis. 2015 Jun;65(6):870-7. doi: 10.1053/j.ajkd.2014.10.017. Epub 2014 Dec 18. PMID 25533599